CLINICAL TRIAL: NCT03719261
Title: Assessment of Postoperative Pain and Antibacterial Activity of Chitosan Nanoparticles Versus Sodium Hypochlorite as a Root Canal Irrigant in Infected Root Canal
Brief Title: Assessment of Pain and Antibacterial Activity of Chitosan Versus Sodium Hypochlorite as Irrigant in Infected Canal
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sarah mahgoub, phD student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sarah mahgoub
Record Dates: First submitted 2018-10-20; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Chitosan; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded The patient is also outcome assessor will be blinded as well as data analyst person.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium hypochlorite (Active Comparator): Sodium hypochlorite (NaOCL) is the most recommended irrigant due to its broad antibacterial effect, necrotic tissues and dentin collagen dissolving capability and inactivation of endotoxins.10ml of 2.5%NaOCL will be used during instrumentation in control group
  Interventions: Drug: Sodium Hypochlorite
- chitosan nanoparticles (Experimental): Chitosan is a bioactive polymer obtained from deacetylation of chitin and is used in biomedical application due to its antimicrobial properties and biocompatibility and ability to resist aging for longer periods provide antibacterial effect in root canal disinfection.10ml of cs-np will be used during instrumentation in intervention group
  Interventions: Drug: chitosan nanoparticles

INTERVENTIONS:
Drug: chitosan nanoparticles — Chitosan is a bioactive polymer obtained from deacetylation of chitin and is used in biomedical application due to its antimicrobial properties and biocompatibility and ability to resist aging for longer periods provide antibacterial effect in root canal disinfection.10ml of cs-np will be used during instrumentation in intervention group
  Other Names: chitosan
  Arms: chitosan nanoparticles
Drug: Sodium Hypochlorite — Sodium hypochlorite (NaOCL) is the most recommended irrigant due to its broad antibacterial effect, necrotic tissues and dentin collagen dissolving capability and inactivation of endotoxins.10ml of 2.5%NaOCL will be used during instrumentation in control group
  Arms: sodium hypochlorite

SUMMARY:
A randomized clinical trial that aims to study the effect of chitosan nanoparticles (CS-np) versus sodium hypochlorite as a root canal irrigant on postoperative pain and antibacterial activity against E.faecalis in infected root canal.

DETAILED DESCRIPTION:
This trial aims to study the effect of chitosan nanoparticles (CS-np) versus sodium hypochlorite as a root canal irrigant on postoperative pain and antibacterial activity against E.faecalis in infected root canal. initial pre-treatment root canal sample will be taken.These will be designated as sample no.1. after first sample, according to random sequence, the patients will be randomly assigned into two groups. In Group I: Sodium hypochlorite (NaOCL 2.5%) will be used during instrumentation of the canals.In Group II: chitosan nanoparticles (CS-np) will be used. after preparation, the sample no.2 will be taken.Pain will be assessed by giving the patient the numerical pain rating scale (NRS) to assess his pain at 24, 48 and 72 hours after the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Young adult Patients, both genders, aging from 18-45 years.
* Patients with permanent mature teeth (closed apex).
* Single rooted single canal necrotic anterior teeth without apical periodontitis or with slight widening of peridontium.
* Patients should be free from any systemic disease.
* Patients with normal periodontal depth less or equal 3 mm.
* Patients who will agree to the consent and will commit to follow-up.

Exclusion Criteria:

* Patients with permanent immature teeth.
* Teeth with vital pulps.
* Patients with facial swelling or acute infection or pain on percussion
* Patients with fistula.
* Teeth with vertical root fractures, internal or external root resorption and calcification
* Teeth with periodontal involvement or periapical bone loss.
* Patients with any systemic disease that may affect predictable outcome.
* Pregnant or lactating females.
* Non-restorable teeth.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
antibacterial activity | two samples will be taken at the same visit of endodontic treatment at day 1, the outcome measures will be assessed after 24h. the data will be reported after study compeletion about 1 year
  antibacterial activity will be evaluated by Sampling and culture method. The samples will be subjected to microbiological analysis to ascertain their individual microbiological load after 24h, this will be analyzed by counting the colony forming units (CFUs).

IPD SHARING:
Plan to Share IPD: No
there is no plan to make the individual participant data available to other researchers.